CLINICAL TRIAL: NCT03500926
Title: Randomized Controlled Trial Comparing a Short Uncemented Femoral Stem to a Similar Standard Uncemented Femoral Stem
Brief Title: Comparison of a Short Uncemented Femoral Stem to a Similar Standard Uncemented Femoral Stem
Acronym: hype
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association pour le Développement et l'Enseignement de la Chirurgie Réparatrice et Orthopédique (Other)
Responsible Party: Principal Investigator, Dr David BIAU, Professor, Association pour le Développement et l'Enseignement de la Chirurgie Réparatrice et Orthopédique
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-A03215-48
Record Dates: First submitted 2018-03-09; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-03

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: randomized 1/1 comparison
Who Masked: Participant
Masking Description: implant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hype standard (Active Comparator): total hip replacement with standard femoral stem
  Interventions: Device: total hip replacement - standard femoral stem
- hype mini (Experimental): total hip replacement with short uncemented femoral stem
  Interventions: Device: total hip replacement - short femoral stem

INTERVENTIONS:
Device: total hip replacement - standard femoral stem — total hip replacement with standard femoral stem
  Arms: hype standard
Device: total hip replacement - short femoral stem — total hip replacement with short femoral stem
  Arms: hype mini

SUMMARY:
This randomized controlled trial will compare patients receiving a standard uncemented femoral stem with patients receiving an identically designed short uncemented femoral stem.

DETAILED DESCRIPTION:
This randomized controlled trial will compare patients receiving a standard uncemented femoral stem with patients receiving an identically designed short uncemented femoral stem.

Patients will be randomized a few days before the operation. At the time of surgery, the surgeon will use the relevant implant. Patients will be followed up for 5 years after surgery. The main outcome criteria is the stem subsidence measured radiographically with a dedicated software.

ELIGIBILITY:
Inclusion Criteria:

* hip osteoarthritis requiring a total hip replacement
* >18 years old
* agrees to participate

Exclusion Criteria:

* total hip replacement not indicated
* general anesthesia contraindicated
* previous surgery on the ipsilateral femur
* follow-up not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-03-09 (Actual); Primary Completion 2022-03-09 (Estimated); Study Completion 2025-03-09 (Estimated)

PRIMARY OUTCOMES:
stem subsidence | 2 years postop
  stem subsidence will be measured using the EBRA (Ein-Bild-Rontgen-analyse) software on postoperative antero-posterior radiographs (5 xrays from day one to year 2)

SECONDARY OUTCOMES:
Intraoperative surgeon satisfaction | intraoperative
  measurement of surgeon's satisfaction with using the instrumentation to insert the stem; on a Likert scale intraoperative complication

OTHER OUTCOMES:
intraoperative proportion of patients requiring a blood transfusion | at time of hospital discharge, at approximately 2 days
  proportion of patients requiring a blood transfusion during the procedure
postoperative PMA (Postel Merle d'Aubigné) score after hospital discharge | 3 months, 1 year, 2 years, 5 years
  PMA score
postoperative Oxford hip score after hospital discharge | 3 months, 1 year, 2 years, 5 years
  oxford hip score
scar assessement | 3 months, 1 year, 2 years, 5 years
  patient specific index
hip pain | 3 months, 1 year, 2 years, 5 years
  measurement of hip pain on a Likert scale
thigh pain | 3 months, 1 year, 2 years, 5 years
  measurement of thigh pain on a Likert scale
revision of hip replacement | at 5 years
  cumulative incidence of revision at 5 years (Cox model)
radiological outcome - engh score | 2 years
  Engh score
radiological outcome - ARA (AGORA Roentgenographic Assessment) score | 2 years
  ARA score
in hospital morphine consumption | postop day 1
  total dose of morphine used in recovery room and until day one
in hospital blood transfusion | until discharge from hospital, at approximately 2 days
  proportion of patients requiring a blood transfusion during hospitalisation
duration of hospital stay | until discharge from hospital, at approximately 2 days
  length of hospitalisation in days

CONTACTS AND LOCATIONS:
Overall Officials: David BIAU, MD, Principal Investigator — Association pour le Développement et l'Enseignement de la Chirurgie Réparatrice et Orthopédique
Locations (1):
- Hopital Cochin, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided